CLINICAL TRIAL: NCT04281979
Title: An MRI Study of Neural Activity Following Exposure to a Specific Substance in Young Cigarette Smokers
Brief Title: Effects of a Specific Substance in Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Angelica Morales, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00018483; K01DA046649 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Smoking
Keywords: Nondaily Smoking; Craving; Impulsivity
MeSH Terms: conditions — Smoking; Impulsive Behavior | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: This study will examine the acute effects of a substance (e.g. stimulant, sedative, analgesic) on a single group of nondaily smokers. All participants will complete 2 experimental sessions under the influence of a substance or placebo. The order of the active and placebo sessions will be randomized.
Who Masked: Participant
Masking Description: In each of the two conditions, participants will be asked to consume a drink and pill. They will be informed that the drink and pill may contain a variety of over the counter substances but they will not be informed about the contents of the drinks and pills until they have completed both the active and placebo visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Agent (Experimental)
  Interventions: Drug: Study Agent
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Study Agent — The study agent will be administered via beverages and/or a capsule. The substances used in the study are legal, non-prescription, and are proven safe for human consumption at the doses used. The study agent may be a depressant (such as alcohol), a stimulant (such as caffeine), or an analgesic (such as aspirin).
  Arms: Study Agent
Drug: Placebo — In the placebo conditions participants will consume beverages and capsules that contain no or very small quantities of the study agent.
  Arms: Placebo

SUMMARY:
Although rates of cigarette use are declining, the proportion of nondaily smokers is rising, particularly among young adults. Among young adults, nondaily smoking is associated with negative health consequences and, for some, may lead to the establishment of life-long smoking patterns. The goal of this project is to understand the behavioral, psychological and neurobiological factors that contribute to cigarette use in nondaily smokers to aid the development of tailored evidence-based interventions.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the neurobiological mechanisms associated with cigarette use in young nondaily smokers (ages 21-25). Nondaily smokers experience fewer symptoms of cigarette withdrawal than daily smokers; however, they still experience difficulty quitting. Since smoking cessation before the age of 30 substantially attenuates the long-term health consequences associated with smoking, understanding the factors that motivate cigarette use in young nondaily smokers and developing tailored interventions will be critical for curbing cigarette use and improving public health. The proposed project will use functional magnetic resonance imaging (fMRI) to examine how other substances (e.g. stimulates, sedatives, or analgesics) impact brain function and will assess the extent to which substance-induced changes in brain function correlate with impulsive choice, cigarette craving, and craving regulation in young adults. Furthermore, the investigators will assess how substance-induced changes in brain function, impulsivity, craving, and capacity for craving regulation predict cigarette use over the course of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 21-40 years old
* Right-handed
* Fluent in English
* Report smoking cigarettes or e-cigarettes 1-27 days in the past month
* Report binge drinking based on NIAAA criteria (5 or more drinks per occasion for males, 4 or more drinks per occasion for females) at least 1 time in the past 90 days without adverse incident

Exclusion Criteria:

* Seeking treatment for substance use (e.g. nicotine or alcohol use)
* Moderate or Severe Nicotine Dependence
* Current alcohol use disorder
* Illicit substance use other than marijuana use in the past year
* Marijuana use more than 10 times in the past year
* Major neurological or medical illness - Significant head trauma - Current use of medication affecting the central nervous system
* MRI contraindications (e.g. irremovable metal on the body or pregnancy)

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Impulsivity | Immediately after beverage/capsule consumption
  Impulsivity will be measured by assessing behavior on a temporal discounting task.
Resting State Functional Connectivity | 35 minutes after beverage/capsule consumption
  Brain function will be measured while participants are resting using functional magnetic resonance imaging
Cigarette Craving and Associated Brain Activation | 50 minutes after beverage/capsule consumption
  Brain function will be measured using functional magnetic resonance imaging while participants complete a Craving Regulation Task
Symptoms of Cigarette Dependence | 1 year follow-up from baseline
  The Fagerström Test of Nicotine Dependence total score will be used to measure changes in cigarette dependence

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to users
Time Frame: After data are published
Access Criteria: Data Use Agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to deleting the data after analyses are completed.